CLINICAL TRIAL: NCT03782454
Title: Quantification of Bacterial DNA in Septic Intensive Care Patients in Relation to Concentration of Antibiotics and Clinical Outcome: A Prospective Observation Study
Brief Title: Quantification of Bacterial DNA in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: JS008
Record Dates: First submitted 2018-12-04; First posted 2018-12-20 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-12

CONDITIONS: Septic Shock; Sepsis Bacterial; Sepsis
Keywords: Bacterial DNA clearance; Droplet digital PCR; Betalactam antibiotics; Acute gastrointestinal index; Cytokines
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intensive care patients with sepsis: Adult patients with verified or suspected sepsis admitted to the intensive care department from the emergency department
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood samples taken every third hour during the first 48 hours of intensive care

SUMMARY:
The purpose of this study is to evaluate whether bacterial DNA clearance measured with droplet digital Polymerase Chain Reaction (ddPCR) can be used as a measure of bacterial load in septic intensive care patients. Furthermore, the aim is to examine a possible relation between clearance of bacterial DNA and clinical outcome in the septic patient, and the relationship between concentration of beta-lactam antibiotics and the clearance of bacterial DNA.

DETAILED DESCRIPTION:
Septic syndrome caused by bloodstream infections represents a major healthcare problem worldwide and is the leading cause of mortality in the non-cardiac intensive care unit (ICU). Despite ongoing research efforts in sepsis, the mortality remains as high as 12-30%.

In severe sepsis, the time to adequate antibiotic therapy has been clearly linked to survival. However, in the emergency room, it is challenging to identify the cause behind the clinical presentation and identify patients who would benefit the most from antibiotic treatment. An indiscriminate use of antibiotics inevitably leads to bacterial resistance and unacceptable adverse events. Thus, there is a great and unmet medical need to develop novel diagnostic instruments that could inform the clinician about who would need antibiotics and who would not benefit from it. Furthermore, early identification of the causal microorganism and the inflammatory status of the patients would improve decisions about treatments and reduce administration of antibiotics.

Today the gold standard for diagnosis of bloodstream infections (BSI) is blood culture followed by identification of species and resistance pattern by standard laboratory procedures. This procedure is associated with a high specificity but also with a low sensitivity. Probable reasons for a negative blood culture despite a strong clinical suspicion could be insufficient blood volume in the culture bottles or antibiotic treatment prior to blood sampling with a subsequent failure of the bacteria to grow in the bottles.

In recent years Polymerase Chain reaction (PCR) has been proposed as a method to determine bacterial DNA based on amplification of specific subunits (16S and 18S) of bacterial ribosomal RNA. PCR require very small amount of DNA. Another advantage is the possibility to determine bacterial species from non-viable bacteria by multiplex PCRs. However most of those multiplex PCRs have shown a limited sensitivity even though they also found clinical relevant pathogens that were not detected with blood cultures. Another limitation is that multiplex-PCR only detects at maximum 95% of all sepsis causing pathogens. In a recent published study the author concluded that a tested multiplex PCR "on whole blood specimens" in adjunct to current culture-based methods provided a clinical add-on value. The future role of PCR and other molecular techniques in the clinical setting needs further evaluation.

A new method that could improve the diagnostics of sepsis and also have the possibility to follow the bacterial DNA load during antibiotic treatment is Droplet Digital PCR (ddPCR). This technique enables an absolute quantification of the sepsis causing pathogen targeting either a species specific gene or the 16S ribosomal DNA (rDNA) gene, present in several copies per bacteria. In ddPCR, the sample is divided into about 20.000 water-in-oil droplets, and in all of them the PCR-reaction occurs. Following PCR, each droplet is analyzed to determine the fraction of PCR-positive droplets giving the amount of bacterial DNA in the original sample. The absolute target DNA template concentration can then be calculated, since the size of the droplets is known, and by using Poisson distribution statistics for the correction of more than one positive reaction in the same droplet.

To identify the sepsis causing pathogen sequencing of the 16S rDNA gene or a shotgun metagenomics approach could be used. In the latter, all DNA in a sample is sequenced using Next Generation Sequencing (NGS) and the sepsis causing pathogen can be both detected and aims to be quantified through bioinformatics data analysis.

During the septic course the patient go from vasodilation to vascular leakage and finally a hypotension. This together with added intravenous fluid treatment will increase the distribution volume with an altered pharmacokinetic state for added antibiotics. Furthermore, decreased kidney function is common in ICU patients and augmented creatinine clearance during the acute phase of sepsis is described with increasing frequency. Therefore, it is difficult to anticipate the optimal antibiotic dose for the septic patient. Indeed, it is shown that in a considerable portion of ICU patients an adequate antibiotic exposure is not achieved and this is associated with negative clinical outcome.

A dysregulated host response is a cornerstone of the current understanding of sepsis pathophysiology. Initially during the sepsis course a proinflammatory response is induced by early activation genes, including cytokines associated with inflammation: tumor necrosis factor (TNF), Interleukin-1(IL-1), IL-12 and IL-18. Simultaneously an immune suppression is induced by anti-inflammatory cytokines i.e IL-10 and transforming growth factor. A disrupted homeostasis of the pro- and anti-inflammatory response is suggested to be part of the dysregulated host response in sepsis although clinically available biomarkers for its identification are lacking. Furthermore, the regulatory mediators involved in this process and the association to bacterial clearance during sepsis needs further investigation.

The gastrointestinal tract may be a source of bacteria and a worsening of the septic inflammation in ICU patients, if the epithelial barrier is disrupted. Thus intact gastrointestinal function is critical in severely diseased patients. There are no clinically available biomarkers of gastrointestinal function; however the recently described acute gastrointestinal injury (AGI) score has been shown to correlate with adverse outcome in ICU-patients.

The aim of the study is to investigate whether bacterial DNA in whole blood measured with ddPCR can be used for assessment of bacterial clearance in septic intensive care patients. To do so the investigators will search for a potential association between bacterial DNA clearance and clearance of bacteremia detected by blood cultures.

Further, the aim is to examine a possible relation between clearance of bacterial DNA, biomarkers of dysregulated host response, and clinical outcome in the septic patient. Outcome is measured as: mortality on ICU, mortality <28 days, days in the ICU, change in Sequential Organ Failure Assessment score(SOFA), time in assisted ventilation, lactate clearance, need of vasopressors, and severity of gastrointestinal injury. Further, the aim is to study the relationship between concentration of beta-lactam antibiotics i.e. the minimal inhibitory concentration for the bacteria (T>MIC) detected and the clearance of bacterial DNA. The material collected will also contribute to reveal the relationship between ddPCR and shot gun sequencing in detecting the sepsis causing bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient at the emergency department with verified or suspected sepsis and who is in need of intensive care.
2. Informed Consent by patient or legal representative.
3. Indication for beta-lactam antibiotics

Exclusion Criteria:

1. < 18 years
2. Patients and/or relatives unable to understand study information.
3. Anaphylactic allergy to beta-lactam antibiotics
4. Patients already treated with antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the emergency department
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Bacterial DNA measured by 16S ddPCR | 48 hours
  copies/mL

SECONDARY OUTCOMES:
Concentration of beta-lactam antibiotics | 48 hours
  mg/mL
Lactate clearance | 48 hours
  mmol/L, clearance %
SOFA | ICU stay up to 30 days
  Sequential Organ Failure Assessment score, from 0(normal) to 24(highest organ dysfunction)
Time in assisted ventilation | ICU stay up to 30 days
  hours
Need of vasopressors | ICU stay up to 30 days
  mcg/kg/hour
Days in the ICU | ICU stay up to 30 days
  Days
AGI score | ICU stay up to 30 days
  Acute Gastrointestinal Injury Score 0(normal) to 4(life-threatening GI complications)
ICU mortality | ICU stay up to 30 days
  Occurence of death during ICU stay
28-day mortality | 28 days
  Occurence of death at day 28
Gastrointestinal complications | 28 days
  Occurence of gastrointestinal complications including GI-bleeding, GI-ischemia, pancreatitis and ileus
Intestinal fatty acid binding protein (I-FABP) | 48 hours
  picogram/mL, biomarker of gastrointestinal injury
Citrulline | 48 hours
  nmol/mL, biomarker of gastrointestinal injury
Nuclear DNA | 48 hours
  copies/mL
Cytokines (Th1 and Th2 signature panel) | 48 hours
  pg/ml
Blood cell populations | 48 hours
  Mean fluorescence intensity/ Antibodies/cell. Monocytes, granulocytes, T-cells, and myeloid derived stem cells including surface markers such as PD-1(Programmed cell death protein 1),PD-L1 (Programmed death ligand 1), and HLA-DR (Human leukocyte Antigen - DR isotype)
HLA-DR messenger RNA (mRNA) | 48 hours
  ratio/reference gene
Procalcitonin | 48 hours
  mcg/L
MicroRNA (miRNA) | 48 hours
  Relative expression/ratio reference gene, transcriptomic and quantitative PCR based measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jan Källman, PhD, Principal Investigator — Region Örebro County; Hans Hjelmqvist, Phd, Principal Investigator — Region Örebro County
Locations (1):
- University Hospital in Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided